CLINICAL TRIAL: NCT01370616
Title: A Phase III, Randomized, Double-Blind, Active Comparator-Controlled Clinical Trial to Study the Efficacy and Safety of Ertapenem Sodium (MK-0826) Versus Piperacillin/Tazobactam Sodium in the Treatment of Diabetic Foot Infections in Chinese Adults
Brief Title: Ertapenem Sodium (MK-0826) Versus Piperacillin/Tazobactam Sodium for the Treatment of Diabetic Foot Infections in Chinese Adults (MK-0826-061)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0826-061
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Infection; Diabetic Foot
Keywords: Infection; Diabetes complications; Diabetes wound infection; Soft tissue infection; Osteomyelitis; Diabetes mellitus
MeSH Terms: conditions — Infections; Diabetic Foot; Diabetes Complications; Soft Tissue Infections; Osteomyelitis; Diabetes Mellitus | interventions — Ertapenem; L 749345; Piperacillin; Tazobactam; Piperacillin, Tazobactam Drug Combination; Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ertapenem sodium (Experimental): Participants received 1.0 g intravenous (IV) ertapenem sodium as a single daily dose at Hour 0 infused over a 30-minute interval , and IV piperacillin/tazobactam-matching placebo at Hours 8 and 16 infused over a 30-minute interval, for 5 to 28 days. Participants may be switched to Amoxicillin/clavulunate potassium 625 mg administered orally, twice daily, from Day 6 to Day 28
  Interventions: Drug: Ertapenem sodium; Drug: Piperacillin/tazobactam-matching placebo; Drug: Amoxicillin/clavulunate potassium
- Piperacillin/tazobactam sodium (Active Comparator): Participants received 4.5 g IV piperacillin/tazobactam at Hours 0, 8, and 16 infused over a 30-minute interval, for 5 to 28 days. Participants may be switched to Amoxicillin/clavulunate potassium 625 mg administered orally, twice daily, from Day 6 to Day 28
  Interventions: Drug: Piperacillin/tazobactam sodium; Drug: Amoxicillin/clavulunate potassium

INTERVENTIONS:
Drug: Ertapenem sodium — Ertapenem sodium, 1.0 g IV daily over 30 minutes at Hour 0 for 5 to 28 days
  Other Names: MK-0826, INVANZ™
  Arms: Ertapenem sodium
Drug: Piperacillin/tazobactam sodium — Piperacillin/tazobactam sodium, 4.5 g, IV every 8 hours, given over 30 minutes at Hours 0, 8, and 16 for 5 to 28 days
  Other Names: Tazocin™
  Arms: Piperacillin/tazobactam sodium
Drug: Piperacillin/tazobactam-matching placebo — Placebo, IV over 30 minutes, 2 times per day at Hours 8 and 16 for 5 to 28 days
  Arms: Ertapenem sodium
Drug: Amoxicillin/clavulunate potassium — If clinically indicated, participants may be switched to Amoxicillin/clavulunate potassium 625 mg administered orally, twice daily, from Day 6 to Day 28

SUMMARY:
This study compared ertapenem sodium to piperacillin/tazobactam sodium for the treatment of moderate to severe diabetic foot infections. The primary hypothesis was that treatment with ertapenem sodium is non-inferior to treatment with piperacillin/tazobactam sodium, in achieving clinical improvement or cure.

ELIGIBILITY:
Inclusion Criteria:

Participant is Chinese with:

* Type I diabetes mellitus (IDDM) or Type II diabetes mellitus (NIDDM) treated with diet and/or medication
* Clinically- or bacteriologically-documented moderate-to-severe (non life-threatening) diabetic foot infection that requires treatment with IV antibiotics
* Wound site or lesion with purulent drainage from the primary site of infection OR at least 3 of the following: fever, white blood count (WBC) >10,000 with >5% immature neutrophils, local periwound erythema (redness) extending >1 cm away from the wound edge or abscess cavity, localized periwound edema (swelling), localized tenderness or pain, localized fluctuance, lymphangitis associated with a skin lesion, localized warmth, and localized induration (limb brawny edema)
* Negative skin test result for allergy to penicillin

Exclusion Criteria:

* Pregnant, breastfeeding, or intending to become pregnant or father a child during the course of the study
* Presence of uncomplicated skin infection such as the following: simple abscesses, impetigo, furunculosis, carbunculosis, or folliculitis in normal hosts; infected burn wound; necrotizing fasciitis; suspected osteomyelitis contiguous with the skin or skin structure infection for which removal of the infected bone is not likely to occur within 2 days of initiation of IV study therapy; wound infection that contains concomitant gangrene that cannot be adequately removed with debridement; infection likely to require a below-the-knee amputation (BKA); infection involving prosthetic material; or evidence of indwelling foreign material (such as prosthetic or surgical hardware) near the infected site that cannot be removed by surgical debridement
* Treatment within 3 days prior to the eligibility screening with >24 hours of systemic antibiotic therapy known to be effective against the presumed or documented etiologic pathogen(s)
* History of serious allergy, hypersensitivity (e.g., anaphylaxis), or any serious reaction to carbapenem antibiotics (such as ertapenem sodium, imipenem cilastatin, meropenem, or doripenem) piperacillin/tazobactam sodium, amoxicillin/clavulanate, any penicillins, any cephalosporins, or any other β-lactam agents
* Need for concomitant systemic antibacterial(s) in addition to those designated in the 2 study groups (with the exception of the addition of vancomycin for Enterococcus ssp. or methicillin-resistant Staphylococcus aureus [MRSA])
* Insufficient vascular perfusion to the affected limb
* Rapidly progressive or terminal illness
* Requirement or anticipation of need for dialysis (peritoneal dialysis, hemodialysis, or hemofiltration)
* Acute hepatitis or acute decompensation of chronic hepatitis
* Human immunodeficiency virus (HIV)-positive with a clinical diagnosis of acquired immune deficiency syndrome (AIDS), or an absolute neutrophil count (ANC) of <1000 cells/mm^3
* Immunosuppression
* Participation in any other clinical study involving the administration of an investigational medication within 30 days
* Participation in any other clinical study involving ertapenem sodium (INVANZ™)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2011-09-02 (Actual); Primary Completion 2013-12-08 (Actual); Study Completion 2013-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Xu ZR, Ran XW, Xian Y, Yan XD, Yuan GY, Mu SM, Shen JF, Zhang BS, Gan WJ, Wang J. Ertapenem versus piperacillin/tazobactam for diabetic foot infections in China: a Phase 3, multicentre, randomized, double-blind, active-controlled, non-inferiority trial. J Antimicrob Chemother. 2016 Jun;71(6):1688-96. doi: 10.1093/jac/dkw004. Epub 2016 Feb 16. PMID 26888908
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0826-061&kw=0826-061&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ertapenem Sodium | Piperacillin/Tazobactam Sodium
Started | 282 (Participants randomized) | 283 (Participants randomized)
Treated | 275 | 275
Completed | 220 | 216
Not Completed | 62 | 67
Not completed — Adverse Event | 11 | 16
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 6 | 2
Not completed — Lost to Follow-up | 0 | 3
Not completed — Physician Decision | 6 | 6
Not completed — Progressive Disease | 0 | 1
Not completed — Recovery | 1 | 0
Not completed — Technical Problems | 3 | 5
Not completed — Withdrawal by Subject | 34 | 34

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Ertapenem Sodium: Participants received 1.0 g IV ertapenem sodium as a single daily dose at Hour 0 infused over a 30-minute interval , and IV piperacillin/tazobactam-matching placebo at Hours 8 and 16 infused over a 30-minute interval, for 5 to 28 days. Participants may be switched to Amoxicillin/clavulunate potassium 625 mg administered orally, twice daily, from Day 6 to Day 28
- Total: Total of all reporting groups
Arm/Group | Ertapenem Sodium | Piperacillin/Tazobactam Sodium | Total
Number analyzed (Participants) | 282 | 283 | 565
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (10.9) | 60.4 (10.1) | 60.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 100 | 201
  Male | 181 | 183 | 364

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Favorable Clinical Response Assessments at Discontinuation of Intravenous (IV) Study Therapy (DCIV)
Description: The investigator assessed participants for a favorable clinical response, defined as clinical improvement or cure. Clinical improvement means that most pretherapy signs and symptoms of the index infection, in particular fever, lympangitis, and purulent drainage had resolved, and no further IV antibiotic therapy was required. Cure means that all pretherapy signs and symptoms of the index infection had resolved, and no further IV antibiotic therapy was required.
Time Frame: Day 5 up to Day 28
Population: Participants with confirmed clinical diagnosis, adequate IV study therapy, protocol-specified visit at DCIV, and no protocol-specific exclusions. A modified last-observation-carried-forward (LOCF), where only failure was carried forward, was used to impute missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ertapenem Sodium | Piperacillin/Tazobactam Sodium
Number analyzed (Participants) | 219 | 224
Percentage of participants | 93.6 [89.5 to 96.5] | 97.3 [94.3 to 99.0]
Statistical Analysis 1: Comparison: Ertapenem Sodium vs Piperacillin/Tazobactam Sodium; Test type: Non-Inferiority or Equivalence — If the 95% confidence interval for the estimated difference between the two groups has a lower bound greater than -15%, then ertapenem sodium will be considered at least as effective as piperacillin/tazobactam sodium; Estimated Difference = -3.8, 95% CI 2-sided [-8.3 to 0.0] — Ertapenem minus Piperacillin/tazobactam. Based on Miettinen & Nurminen method stratified by the severity of diabetes foot infection

2. Secondary Outcome: Percentage of Participants With Favorable Clinical Response Assessments at Day 5 of IV Study Therapy
Description: as for outcome 1
Time Frame: Day 5
Population: Participants with a confirmed clinical diagnosis, adequate length of IV study therapy, protocol-specified visit at Day 5, and no documented protocol-specific exclusions. A modified LOCF, where only failure was carried forward, was used to impute missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ertapenem Sodium | Piperacillin/Tazobactam Sodium
Number analyzed (Participants) | 210 | 221
Percentage of participants | 96.2 [92.6 to 98.3] | 97.7 [94.8 to 99.3]
Statistical Analysis 1: Comparison: Ertapenem Sodium vs Piperacillin/Tazobactam Sodium; Test type: Superiority or Other; Estimated Difference = -1.7, 95% CI 2-sided [-5.5 to 1.8] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With Favorable Clinical Response Assessments at Follow-up Assessment (FUA) Day 10 of Post-antibiotic Study Therapy
Description: as for outcome 1
Time Frame: Day 15 up to Day 38
Population: Participants with a confirmed clinical diagnosis, adequate length of IV study therapy, protocol-specified visit at FUA, and no documented protocol-specific exclusions. A modified LOCF, where only failure was carried forward, was used to impute missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ertapenem Sodium | Piperacillin/Tazobactam Sodium
Number analyzed (Participants) | 193 | 195
Percentage of participants | 92.2 [87.5 to 95.6] | 94.4 [90.1 to 97.2]
Statistical Analysis 1: Comparison: Ertapenem Sodium vs Piperacillin/Tazobactam Sodium; Test type: Superiority or Other; Estimated Difference = -2.3, 95% CI 2-sided [-7.7 to 2.8] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants With Favorable Microbiological Response Assessments at FUA Day 10 of Post-antibiotic Study Therapy
Description: The investigator assessed participants for a favorable microbiological response, defined as eradication or presumptive eradication. Eradication means that the original pathogen was absent from the last available culture of an adequate specimen obtained from the original site of infection. Presumptive eradication means that the participant showed cure or improvement and no appropriate material is available to follow-up culture from the original site of infection, or collection of such a specimen would cause undue discomfort.
Time Frame: Day 15 up to Day 38
Population: Participants with proper clinical diagnosis, adequate study therapy, adequate clinical assessment, appropriate antimicrobial therapy, and proper microbiological assessment. A modified LOCF, where only failure was carried forward, was used to impute missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ertapenem Sodium | Piperacillin/Tazobactam Sodium
Number analyzed (Participants) | 140 | 149
Percentage of participants | 86.4 [79.6 to 91.6] | 89.9 [83.9 to 94.3]
Statistical Analysis 1: Comparison: Ertapenem Sodium vs Piperacillin/Tazobactam Sodium; Test type: Superiority or Other; Estimated Difference = -4.1, 95% CI 2-sided [-11.9 to 3.4] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With Both Favorable Clinical and Microbiological Response Assessments at FUA Day 10 of Post-antibiotic Study Therapy
Description: The investigator assessed participants for both a favorable clinical response (clinical improvement or cure) and a favorable microbiological response (eradication or presumptive eradication). Clinical improvement means that most pretherapy signs and symptoms of the index infection, had resolved, and no further IV antibiotic therapy is required. Cure means that all pretherapy signs and symptoms of the index infection had resolved, and no further IV antibiotic therapy was required. Eradication means that the original pathogen was absent from the last available culture obtained from the original site of infection. Presumptive eradication means that the participant showed cure or improvement and no appropriate material is available to follow-up culture from the original site of infection, or collection of such a specimen would cause undue discomfort.
Time Frame: Day 15 up to Day 38
Population: Participants with proper clinical diagnosis, adequate study therapy and clinical assessment, appropriate antimicrobial therapy, and microbiological assessment. One participant from the Ertapenem arm with indeterminate clinical response, was excluded from the analysis. A modified LOCF (failure was carried forward), was used to impute missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ertapenem Sodium | Piperacillin/Tazobactam Sodium
Number analyzed (Participants) | 139 | 149
Percentage of participants | 86.3 [79.5 to 91.6] | 89.9 [83.9 to 94.3]
Statistical Analysis 1: Comparison: Ertapenem Sodium vs Piperacillin/Tazobactam Sodium; Test type: Superiority or Other; Estimated Difference = -4.3, 95% CI 2-sided [-12.1 to 3.3] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants With One or More Adverse Events (AEs)
Description: An AE is any unfavorable and unintended change in the structure, function, or chemistry of the body that is temporally associated with the use of the investigational product, whether or not considered related to the use of the medicinal product. This also includes any change in frequency and/or intensity of a preexisting condition which is temporally associated with the use of the medicinal product.
Time Frame: Up to day 42
Population: Participants who received at least one dose of IV study therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Ertapenem Sodium | Piperacillin/Tazobactam Sodium
Number analyzed (Participants) | 275 | 275
Percentage of participants | 64.0 | 56.7
Statistical Analysis 1: Comparison: Ertapenem Sodium vs Piperacillin/Tazobactam Sodium; Test type: Superiority or Other; Estimated Difference = 7.3, 95% CI 2-sided [-0.9 to 15.4] — Ertapenem minus Piperacillin/tazobactam group. Based on Miettinen & Nurminen method without adjusting strata

7. Secondary Outcome: Percentage of Participants With Drug-related AEs
Description: A drug-related AE is any AE caused by the test drug as determined by an investigator who is a qualified physician. Drug-relatedness of the AE was assessed by evidence that the participant was actually exposed to the test drug, whether the AE followed a reasonable temporal sequence from administration of the test drug, and whether or not the AE was more reasonably explained by another source.
Time Frame: Up to day 42
Population: Participants who received at least one dose of IV study therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Ertapenem Sodium | Piperacillin/Tazobactam Sodium
Number analyzed (Participants) | 275 | 275
Percentage of participants | 13.5 | 16.0
Statistical Analysis 1: Comparison: Ertapenem Sodium vs Piperacillin/Tazobactam Sodium; Test type: Superiority or Other; Estimated Difference = -2.5, 95% CI 2-sided [-8.5 to 3.4] — Ertapenem minus Piperacillin/tazobactam group. Based on Miettinen & Nurminen method without adjusting strata

8. Secondary Outcome: Percentage of Participants With Serious AEs (SAEs)
Description: A SAE is an AE occurring at any dose that resulted in any of the following: death, was life threatening, a persistent or significant disability/incapacity, prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect in an offspring, was a cancer, an overdose, or other important medical events requiring medical or surgical intervention.
Time Frame: Up to day 42
Population: Participants who received at least one dose of IV study therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Ertapenem Sodium | Piperacillin/Tazobactam Sodium
Number analyzed (Participants) | 275 | 275
Percentage of participants | 6.2 | 4.4
Statistical Analysis 1: Comparison: Ertapenem Sodium vs Piperacillin/Tazobactam Sodium; Test type: Superiority or Other; Estimated Difference = 1.8, 95% CI 2-sided [-2.0 to 5.8] — Ertapenem minus Piperacillin/tazobactam group. Based on Miettinen & Nurminen method without adjusting strata

9. Secondary Outcome: Percentage of Participants Who Discontinued Treatment Due to an AE
Description: Participants chose to discontinue treatment or were discontinued from the study by the investigator due to any untoward effects, or for safety reasons such as an AE. The investigator determined whether or not the AE caused the test drug to be discontinued.
Time Frame: Up to day 28
Population: Participants who received at least one dose of IV study therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Ertapenem Sodium | Piperacillin/Tazobactam Sodium
Number analyzed (Participants) | 275 | 275
Percentage of participants | 4.0 | 5.8
Statistical Analysis 1: Comparison: Ertapenem Sodium vs Piperacillin/Tazobactam Sodium; Test type: Superiority or Other; Estimated Difference = -1.8, 95% CI 2-sided [-5.7 to 1.9] — Ertapenem minus Piperacillin/tazobactam group. Based on Miettinen & Nurminen method without adjusting strata

ADVERSE EVENTS:
Time Frame: Through 14-Day follow-up (up to Day 42)
Description: Participants who received at least one dose of IV study therapy
Arm/Group | Ertapenem Sodium | Piperacillin/Tazobactam Sodium
Serious Adverse Events (participants affected / at risk) | 17/275 | 12/275
Other Adverse Events (participants affected / at risk) | 102/275 | 89/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertapenem Sodium (N=275) | Piperacillin/Tazobactam Sodium (N=275)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Choroidal detachment (Eye disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 4 (4) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertapenem Sodium (N=275) | Piperacillin/Tazobactam Sodium (N=275)
Constipation (Gastrointestinal disorders) | 16 (17) | 14 (17)
Diarrhoea (Gastrointestinal disorders) | 16 (17) | 11 (11)
Pyrexia (General disorders) | 21 (27) | 21 (29)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 16 (16)
Alanine aminotransferase increased (Investigations) | 35 (36) | 19 (19)
Aspartate aminotransferase increased (Investigations) | 32 (32) | 19 (19)
Hypoglycaemia (Metabolism and nutrition disorders) | 16 (19) | 16 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (13) | 16 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.